CLINICAL TRIAL: NCT01212510
Title: Study of Circulating Markers in Serum of Patients Treated for Metastatic Colorectal Cancer
Acronym: Coca-Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/170/HP
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; circulating tumor markers; circulating tumor cell; circulating tumor DNA; marker's kinetic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tumor markers (Other): measurement of tumor markers ( blood rate of ACE, CA19-9, circulating tumor cell, circulating tumor DNA )
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — blood rate of ACE, CA19-9, circulating tumor cell, circulating tumor DNA

SUMMARY:
The primary purpose of the study is to confirm the results of previous study about the usefulness of the serum Carcinoembryonic antigen (CEA) kinetic for chemotherapy monitoring in patients with unresectable metastasis of colorectal cancer (J Clin Oncol 2008;26:3681-6). The secondary purpose is to evaluate the value of circulating free mutant DNA and circulating tumor cells (CTC) and their variations during the treatment.

DETAILED DESCRIPTION:
Prospective cohort study of patients treated with systemic chemotherapy for unresectable metastatic colorectal cancer. The chemotherapy monitoring is currently based on radiological evaluation (RECIST criteria) and clinical evaluation. Circulating markers as CEA, free mutant DNA, CTC represent an alternative approach. A previous study on usefulness of the serum Carcinoembryonic antigen (CEA) kinetic for chemotherapy monitoring in patients with unresectable metastasis of colorectal cancer has been published (J Clin Oncol 2008;26:3681-6). The present study is designed to validate the previous data. The secondary purpose is to evaluate variations of free mutant DNA and CTC during the chemotherapy. Patients will be included prospectively in 4 centers in Normandy. All systemic chemotherapy and biotherapy validate in this clinical situation by the French National Cancer Institute (INCa) is accepted. Evaluation of response based on RECIST criteria will be performed every 3 months. Blood samples for CEA and CA 19-9 levels will be performed every courses of chemotherapy during first 3 months. Blood samples for detection of free mutant DNA and CTC will be performed at day 1 and 42 of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has Stage IV colorectal adenocarcinoma histologically proved
* Patient has at least one measurable lesion
* Patient has performance status 0-2 on the WHO performance scale
* Patient is male or female, and > 18 years of age
* Patient has agree to participate by giving written informed consent

Exclusion Criteria:

* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Prediction of tumor progression | 3 months
  sensitivity and specificity of CEA kinetic to predict tumor progression at 3 months (RECIST)

SECONDARY OUTCOMES:
Prediction of tumor response | 3 months
  sensitivity and specificity of CEA kinetic to predict tumor response at 3 months (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MICHEL, Pr, Principal Investigator — UH Rouen
Locations (4):
- France (4):
  - Centre François Baclesse, Caen
  - University Hospital, Caen
  - Centre Frédéric Joliot, Rouen
  - University Hospital, Rouen

REFERENCES:
- [Derived] Sefrioui D, Beaussire L, Gillibert A, Blanchard F, Toure E, Bazille C, Perdrix A, Ziegler F, Gangloff A, Hassine M, Elie C, Bignon AL, Parzy A, Gomez P, Thill C, Clatot F, Sabourin JC, Frebourg T, Benichou J, Bouhier-Leporrier K, Gallais MP, Sarafan-Vasseur N, Michel P, Di Fiore F. CEA, CA19-9, circulating DNA and circulating tumour cell kinetics in patients treated for metastatic colorectal cancer (mCRC). Br J Cancer. 2021 Aug;125(5):725-733. doi: 10.1038/s41416-021-01431-9. Epub 2021 Jun 10. PMID 34112948